CLINICAL TRIAL: NCT01942707
Title: Study of Scarpa´s Fascia in the Formation of Seroma Post Abdominoplasty After Bariatric Surgery
Brief Title: Scarpa´s Fascia in the Formation of Seroma Post Abdominoplasty After Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Heraldo Carlos Borges, M D - Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: INFORZATO55
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Seroma
Keywords: Abdominoplasty,Seroma,Bariatric surgery
MeSH Terms: conditions — Seroma | interventions — Abdominoplasty

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient will not know if the Scarpa´s fascia has been removed or preserved.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abdominoplasty without Scarpa´s Facia (Active Comparator): Anchor-line abdominoplasty where the Scarpa's Fascia will be removed.
  Interventions: Procedure: Abdominoplasty without Scarpa´s Facia
- abdominoplasty with Scarpa's Fascia (Experimental): Anchor-line abdominoplasty where the Scarpa's Fascia will be preserved.
  Interventions: Procedure: abdominoplasty with Scarpa's Fascia

INTERVENTIONS:
Procedure: abdominoplasty with Scarpa's Fascia — During surgical detachment of the abdominal flap the Scarpa´s fascia is preserved.
  Arms: abdominoplasty with Scarpa's Fascia
Procedure: Abdominoplasty without Scarpa´s Facia — During surgical detachment of the abdominal flap the Scarpa´s fascia is removed.
  Arms: Abdominoplasty without Scarpa´s Facia

SUMMARY:
46 female postbariatric patients will be submitted to anchor-line abdominoplasty with drains insertion. Patients will be randomized to two groups. One group will have the Fascia Scarpa removed and in the other the Fascia Scarpa will be preserved. The drains will be removed when the volume is less than 30 ml in 24 hours. The primary outcome will be the volume of total drainage obtained in the drains of the abdominal region. Secondary outcomes will be the length of time the drains remain and the presence of seroma assessed by ultrasound on the twentieth postoperative day.

DETAILED DESCRIPTION:
Morbid obesity has been increasing in Brazil and the world and bariatric surgery is the most effective and long-lasting treatment. This leads to large weight losses leading to large body deformities due to excess skin and subcutaneous tissue. The most common post-bariatric plastic surgery is post-bariatric abdominoplasty which main complication is seroma. PURPOSE: To evaluate the effect of Scarpa fascia preservation in seroma reduction. METHODS: A total of 46 patients were randomly assigned to two groups. One group will have the Fascia Scarpa removed and in the other the Fascia Scarpa will be preserved. The drains will be removed when the volume is less than 30 ml in 24 hours. The primary outcome will be the volume of total drainage obtained in the drains of the abdominal region. Secondary outcomes will be the length of time the drains remain and the presence of seroma assessed by ultrasound on the twentieth postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 22 and 30 Kg/m2
* Female post-bariatric patient

Exclusion Criteria:

* neoplasms
* Diabetes
* lymphatic system diseases
* abdominal scars except C section and bariatric surgery scars
* mental disorders

Ages: 24 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2013-03; Primary Completion 2018-04 (Estimated); Study Completion 2018-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lydia M Ferreira, MD, Phd, Study Chair — Federal University of São Paulo; Juan C Montano-Pedroso, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrades P, Prado A. Composition of postabdominoplasty seroma. Aesthetic Plast Surg. 2007 Sep-Oct;31(5):514-8. doi: 10.1007/s00266-007-0078-3. Epub 2007 Jul 20. PMID 17659406
- [Background] Andrades P, Prado A, Danilla S, Guerra C, Benitez S, Sepulveda S, Sciarraffia C, De Carolis V. Progressive tension sutures in the prevention of postabdominoplasty seroma: a prospective, randomized, double-blind clinical trial. Plast Reconstr Surg. 2007 Sep 15;120(4):935-946. doi: 10.1097/01.prs.0000253445.76991.de. PMID 17805122
- [Background] Baroudi R, Ferreira CA. Seroma: how to avoid it and how to treat it. Aesthet Surg J. 1998 Nov-Dec;18(6):439-41. doi: 10.1016/s1090-820x(98)70073-1. PMID 19328174
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Bussolaro RA, Garcia EB, Zanella MT, Ferreira LM. Impaired abdominal skin sensory function in morbid obesity and after bariatric surgery. Obes Surg. 2012 Mar;22(3):353-9. doi: 10.1007/s11695-011-0485-z. PMID 21805192
- [Background] Bercial ME, Sabino Neto M, Calil JA, Rossetto LA, Ferreira LM. Suction drains, quilting sutures, and fibrin sealant in the prevention of seroma formation in abdominoplasty: which is the best strategy? Aesthetic Plast Surg. 2012 Apr;36(2):370-3. doi: 10.1007/s00266-011-9807-8. Epub 2011 Aug 20. PMID 21858593
- [Background] Colquitt J, Clegg A, Loveman E, Royle P, Sidhu MK. Surgery for morbid obesity. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD003641. doi: 10.1002/14651858.CD003641.pub2. PMID 16235331
- [Background] Costa LF, Landecker A, Manta AM. Optimizing body contour in massive weight loss patients: the modified vertical abdominoplasty. Plast Reconstr Surg. 2004 Dec;114(7):1917-23; discussion 1924-6. doi: 10.1097/01.prs.0000142997.63346.95. PMID 15577368
- [Background] Dellon AL. Fleur-de-lis abdominoplasty. Aesthetic Plast Surg. 1985;9(1):27-32. doi: 10.1007/BF01570680. PMID 3158172
- [Background] Di Martino M, Nahas FX, Barbosa MVJ, Montecinos Ayaviri NA, Kimura AK, Barella SM, Novo NF, Ferreira LM. Seroma in lipoabdominoplasty and abdominoplasty: a comparative study using ultrasound. Plast Reconstr Surg. 2010 Nov;126(5):1742-1751. doi: 10.1097/PRS.0b013e3181efa6c5. PMID 20639797
- [Background] Costa-Ferreira A, Rebelo M, Vasconez LO, Amarante J. Scarpa fascia preservation during abdominoplasty: a prospective study. Plast Reconstr Surg. 2010 Apr;125(4):1232-1239. doi: 10.1097/PRS.0b013e3181d0ac59. PMID 20072084
- [Background] Farah AB, Nahas FX, Ferreira LM, Mendes Jde A, Juliano Y. Sensibility of the abdomen after abdominoplasty. Plast Reconstr Surg. 2004 Aug;114(2):577-82; discussion 583. doi: 10.1097/01.prs.0000128356.93462.7b. PMID 15277836
- [Background] Fraccalvieri M, Datta G, Bogetti P, Verna G, Pedrale R, Bocchiotti MA, Boriani F, Obbialero FD, Kefalas N, Bruschi S. Abdominoplasty after weight loss in morbidly obese patients: a 4-year clinical experience. Obes Surg. 2007 Oct;17(10):1319-24. doi: 10.1007/s11695-007-9235-7. PMID 18000727
- [Background] Garcia-Garcia ML, Martin-Lorenzo JG, Campillo-Soto A, Torralba-Martinez JA, Liron-Ruiz R, Miguel-Perello J, Mengual-Ballester M, Aguayo-Albasini JL. [Complications and level of satisfaction after dermolipectomy and abdominoplasty post-bariatric surgery]. Cir Esp. 2014 Apr;92(4):254-60. doi: 10.1016/j.ciresp.2013.04.024. Epub 2013 Dec 18. Spanish. PMID 24360407
- [Background] Gloy VL, Briel M, Bhatt DL, Kashyap SR, Schauer PR, Mingrone G, Bucher HC, Nordmann AJ. Bariatric surgery versus non-surgical treatment for obesity: a systematic review and meta-analysis of randomised controlled trials. BMJ. 2013 Oct 22;347:f5934. doi: 10.1136/bmj.f5934. PMID 24149519
- [Background] James PT. Obesity: the worldwide epidemic. Clin Dermatol. 2004 Jul-Aug;22(4):276-80. doi: 10.1016/j.clindermatol.2004.01.010. PMID 15475226
- [Background] Koller M, Hintringer T. Scarpa fascia or rectus fascia in abdominoplasty flap elevation: a prospective clinical trial. Aesthetic Plast Surg. 2012 Apr;36(2):241-3. doi: 10.1007/s00266-011-9795-8. Epub 2011 Aug 19. PMID 21853405
- [Background] Le Louarn C. Partial subfascial abdominoplasty. Aesthetic Plast Surg. 1996 Mar-Apr;20(2):123-7. doi: 10.1007/BF02275530. PMID 8661592
- [Background] Maggard MA, Shugarman LR, Suttorp M, Maglione M, Sugerman HJ, Livingston EH, Nguyen NT, Li Z, Mojica WA, Hilton L, Rhodes S, Morton SC, Shekelle PG. Meta-analysis: surgical treatment of obesity. Ann Intern Med. 2005 Apr 5;142(7):547-59. doi: 10.7326/0003-4819-142-7-200504050-00013. PMID 15809466
- [Background] Mohammad JA, Warnke PH, Stavraky W. Ultrasound in the diagnosis and management of fluid collection complications following abdominoplasty. Ann Plast Surg. 1998 Nov;41(5):498-502. doi: 10.1097/00000637-199811000-00008. PMID 9827952
- [Background] Montano-Pedroso JC, Garcia EB, Omonte IR, Rocha MG, Ferreira LM. Hematological variables and iron status in abdominoplasty after bariatric surgery. Obes Surg. 2013 Jan;23(1):7-16. doi: 10.1007/s11695-012-0720-2. PMID 22820956
- [Background] Nahas FX, Ferreira LM, Ghelfond C. Does quilting suture prevent seroma in abdominoplasty? Plast Reconstr Surg. 2007 Mar;119(3):1060-4; discussion 1065-6. doi: 10.1097/01.prs.0000242493.11655.68. PMID 17312514
- [Background] Nahas FX, di Martino M, Ferreira LM. Fibrin glue as a substitute for quilting suture in abdominoplasty. Plast Reconstr Surg. 2012 Jan;129(1):212e-213e. doi: 10.1097/PRS.0b013e3182365d65. No abstract available. PMID 22186572
- [Background] Neaman KC, Hansen JE. Analysis of complications from abdominoplasty: a review of 206 cases at a university hospital. Ann Plast Surg. 2007 Mar;58(3):292-8. doi: 10.1097/01.sap.0000239806.43438.54. PMID 17471135
- [Background] Persichetti P, Simone P, Scuderi N. Anchor-line abdominoplasty: a comprehensive approach to abdominal wall reconstruction and body contouring. Plast Reconstr Surg. 2005 Jul;116(1):289-94. doi: 10.1097/01.prs.0000170049.94288.d2. PMID 15988280
- [Background] Pitanguy I. Evaluation of body contouring surgery today: a 30-year perspective. Plast Reconstr Surg. 2000 Apr;105(4):1499-514; discussion 1515-6. PMID 10744246
- [Background] Rossetto LA, Garcia EB, Abla LF, Neto MS, Ferreira LM. Quilting suture in the donor site of the transverse rectus abdominis musculocutaneous flap in breast reconstruction. Ann Plast Surg. 2009 Mar;62(3):240-3. doi: 10.1097/SAP.0b013e318180c8e2. PMID 19240517
- [Background] Saldanha OR, Federico R, Daher PF, Malheiros AA, Carneiro PRG, Azevedo SFD, Saldanha Filho OR, Saldanha CB. Lipoabdominoplasty. Plast Reconstr Surg. 2009 Sep;124(3):934-942. doi: 10.1097/PRS.0b013e3181b037e3. PMID 19730314
- [Background] Stewart KJ, Stewart DA, Coghlan B, Harrison DH, Jones BM, Waterhouse N. Complications of 278 consecutive abdominoplasties. J Plast Reconstr Aesthet Surg. 2006;59(11):1152-5. doi: 10.1016/j.bjps.2005.12.060. Epub 2006 Jul 5. PMID 17046623

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment began in october 2014 until april 2015 at Hospital Santo Amaro (private hospital), in Guarujá city, Brazil.
Groups:
- Anchor-line Abdominoplasty Without Scarpa's Fascia: Anchor-line abdominoplasty. The Scarpa's Fascia will be removed in this group.
- Anchor-line Abdominoplasty With Scarpa's Fascia: Anchor-line abdominoplasty. In this group the Scarpa's Fascia will be preserved.
Period: Overall Study
Arm/Group | Anchor-line Abdominoplasty Without Scarpa's Fascia | Anchor-line Abdominoplasty With Scarpa's Fascia
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Keeping Scarpa's Fascia: Abdominoplasty in anchor-line without keeping Scarpa's Fascia.
  Abdominoplasty in anchor-line: Abdominoplasty in anchor-line was performed in both groups
- Keeping Scarpa's Fascia: Abdominoplasty in anchor-line keeping Scarpa's Fascia.
  Abdominoplasty in anchor-line: Abdominoplasty in anchor-line was performed in both groups
- Total: Total of all reporting groups
Arm/Group | No Keeping Scarpa's Fascia | Keeping Scarpa's Fascia | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] — Age as informed by the patient
  years | 37.086 (8.06) | 38.1304 (8.05) | 37.6087 (8.074)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 23 | 23 | 46
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 23 | 23 | 46
BMI [Mean (Standard Deviation); unit: Kg/m2] | 26.4 (3) | 28.2 (1.9) | 27.3 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Total Volume of Drainage in ml.
Description: We will measure the total volume of drainage, in ml, obtained by the drains in the abdominal region. The measure of drainage will be done at the same time (8:00 am) and by the same nurse everyday in all patients until the drain is withdrawn. The drain will be withdrawn when the drained volume is less than 30 ml in 24 hours. Total volume of drainage will be calculated as the sum of the volumes obtained daily.
Time Frame: number of days required for drain withdrawal (drained volume less than 30 ml in 24 hours) and no later than 10 days
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Without Scarpa's Fascia: Abdominoplasty in anchor-line without keeping Scarpa's Fascia.
  Abdominoplasty in anchor-line: Abdominoplasty in anchor-line was performed in both groups
- With Scarpa's Fascia: Abdominoplasty in anchor-line keeping Scarpa's Fascia.
  Abdominoplasty in anchor-line: Abdominoplasty in anchor-line was performed in both groups
Arm/Group | Without Scarpa's Fascia | With Scarpa's Fascia
Number analyzed (Participants) | 23 | 23
ml | 428.9 (222.6) | 249.1 (98.2)
Statistical Analysis 1: Comparison: Without Scarpa's Fascia vs With Scarpa's Fascia; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 179, Standard Deviation 222

2. Secondary Outcome: Number of Days Required for Drain Withdrawal.
Description: Number of days required for drain withdrawal. The measure of drainage will be done at the same time (8:00 am) and by the same nurse everyday in all patients until the drain is withdrawn. The drain will be withdrawn when the drained volume is less than 30 ml in 24 hours.
Time Frame: Number of days required for drain withdrawal (drained volume less than 30 ml in 24 hours) and no later than 10 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Without Scarpa's Fascia | With Scarpa's Fascia
Number analyzed (Participants) | 23 | 23
days | 5.4 (1.9) | 4.2 (1.2)
Statistical Analysis 1: Comparison: Without Scarpa's Fascia vs With Scarpa's Fascia; Test type: Superiority; p = 0.012, t-test, 2 sided; Mean Difference (Final Values) = 1.2, Standard Deviation 1.9

3. Secondary Outcome: Volume of Seroma Assessed by Ultrasound of the Abdominal Wall.
Description: An ultrasound of the abdominal wall will be realized to check the volume of any residual seroma.
Time Frame: Done after 20 days of surgery
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Without Scarpa's Fascia | With Scarpa's Fascia
Number analyzed (Participants) | 23 | 23
ml | 21.6 (40.7) | 16.8 (25)
Statistical Analysis 1: Comparison: Without Scarpa's Fascia vs With Scarpa's Fascia; Test type: Superiority; p = 0.809, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 4.8, Standard Deviation 40.7

ADVERSE EVENTS:
Time Frame: 60 days
Groups:
- Anchor-line Abdominoplasty Without Scarpa's Fascia: Anchor-line Abdominoplasty where the Scarpa's Fascia will be removed.
- Anchor-line Abdominoplasty With Scarpa's Fascia: Anchor-line abdominoplasty where the Scarpa´s Fascia will be preserved.
Arm/Group | Anchor-line Abdominoplasty Without Scarpa's Fascia | Anchor-line Abdominoplasty With Scarpa's Fascia
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT01942707/SAP_000.pdf
  • Study Protocol (2017-10-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT01942707/Prot_001.pdf